CLINICAL TRIAL: NCT00817427
Title: Sleep Disturbance as a Non-Traditional Risk Factor in CKD
Brief Title: Sleep Disturbances as a Risk Factor in Chronic Kidney Disease
Acronym: CRIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: #14075A; 5RO1DK71696-4; 5R01DK071696 (NIH)
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Poor sleep; CKD; Kidney Failure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Baseline (No Intervention): CKD subjects and healthy, matched controls will have measures of cardiovascular function (BP, HR) measure of hormonal fluid balance (renin/aldosterone) measure and measures of glucose metabolism (response to glucose load and over 24 hr profile) with 3 days of habitual sleep time
- CKD- Sleep extension (Experimental): Measures as in baseline but with bed time increased by 2 hours
  Interventions: Other: CKD- sleep extension
- Controls short sleep (Experimental): Measures as in baseline but with sleep disruption
  Interventions: Other: Controls Short sleep

INTERVENTIONS:
Other: Controls Short sleep — Healthy control subject's bedtime will be decreased by 2 hours/night with acoustic sleep disruption
  Other Names: Sleep intervention
  Arms: Controls short sleep
Other: CKD- sleep extension — Sleep will be increased by 2 hours each night for 3 nights
  Other Names: Sleep intervention
  Arms: CKD- Sleep extension

SUMMARY:
This study is designed to determine if either short night time sleep or poor night time sleep could be a risk factor for increasing the rate at which kidney function deteriorates in persons with mild to moderate kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Mild to Moderate CKD
* Healthy controls age and gender matched to CKD subjects
* Regular bedtimes of at least 6h/night, sedentary lifestyle

Exclusion Criteria:

* Diabetes
* Current or previous dialysis for more than 1 month
* Uncontrolled hypertension
* Heart failure
* Liver disease
* HIV
* Hemoglobin < 10.5 g/dl
* Treatment with EProcrit, Epogen, or Aranesp
* Bone or organ transplant,
* Use of immunosuppressive drugs within past 6 months
* Current oral contraceptive use
* Current pregnancy
* Chemotherapy for malignancy within past 2 years

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Comparison of chronobiological profiles of renin/aldosterone, sympatho-vagal balance and CV function in CKD subjects to controls at baseline and after extended sleep in CKD subjects and after decreased time and quality of sleep in control subjects. | Immediately after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Eve Van Cauter, PhD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States